CLINICAL TRIAL: NCT02612311
Title: Phase 3, Randomized Study to Assess the Efficacy and Safety of Ublituximab in Combination With TGR-1202 (Umbralisib) Compared to Obinutuzumab in Combination With Chlorambucil in Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Ublituximab + TGR-1202 Compared to Obinutuzumab + Chlorambucil in Participants With Untreated and Previously Treated Chronic Lymphocytic Leukemia
Acronym: UNITY-CLL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic/Business decision
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTX-TGR-304; 2015-005758-36 (EudraCT Number)
Record Dates: First submitted 2015-11-18; First posted 2015-11-23 (Estimated); Results first posted 2024-05-07 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab; ublituximab; umbralisib; Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Ublituximab + Umbralisib (Experimental): Participants received ublituximab, 150 milligrams (mg), intravenously (IV), on Day 1, 750 mg on Day 2, followed by 900 mg on Days 8 and 15 of Cycle 1 (cycle length=28 days), Day 1 of Cycles 2-6, and once every 3 cycles thereafter, along with umbralisib, 800 mg, orally, once daily during each cycle until disease progression, lack of tolerability, or until the treatment is commercially available or up to 87 months.
  Interventions: Biological: Ublituximab; Drug: TGR-1202
- Arm B: Obinutuzumab + Chlorambucil (Active Comparator): Participants received Obinutuzumab 100 mg, IV on Day 1, 900 mg on Day 2, followed by 1000 mg on Days 8 and 15 of cycle 1 (cycle length = 28 days), Day 1 of Cycle 2-6 along with Chlorambucil 0.5 milligram per kilogram (mg/kg) tablet orally on Days 1 and 15 once daily during each cycle until disease progression, lack of tolerability, or until the treatment is commercially available or up to 87 months.
  Interventions: Biological: Obinutuzumab; Drug: Chlorambucil
- Arm C: Ublituximab (Experimental): Participants received ublituximab, 150 mg, IV, on Day 1, 750 mg on Day 2, followed by 900 mg on Days 8 and 15 of Cycle 1 (cycle length=28 days), Day 1 of Cycles 2-6, and once every 3 cycles thereafter, until disease progression, lack of tolerability, or until the treatment is commercially available or up to 87 months.
  Interventions: Biological: Ublituximab
- Arm D: Umbralisib (Experimental): Participants received umbralisib, 800 mg tablets, orally, once daily during each cycle (cycle length= 28 days) until removal from study or up to 87 months.
  Interventions: Drug: TGR-1202

INTERVENTIONS:
Biological: Obinutuzumab — Obinutuzumab: IV infusion
  Other Names: GAZYVA
  Arms: Arm B: Obinutuzumab + Chlorambucil
Biological: Ublituximab — Ublituximab: IV infusion
  Arms: Arm A: Ublituximab + Umbralisib; Arm C: Ublituximab
Drug: TGR-1202 — TGR-1202: Oral daily dose
  Arms: Arm A: Ublituximab + Umbralisib; Arm D: Umbralisib
Drug: Chlorambucil — Chlorambucil: Oral dose
  Other Names: Leukeran
  Arms: Arm B: Obinutuzumab + Chlorambucil

SUMMARY:
This study evaluates the combination of ublituximab, a novel monoclonal antibody, and TGR-1202, a novel PI3K delta inhibitor compared to obinutuzumab and chlorambucil, and compared to ublituximab or TGR-1202 alone in Chronic Lymphocytic Leukemia (CLL) participants.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve or previously treated Chronic Lymphocytic Leukemia (CLL) requiring treatment
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2

Exclusion Criteria:

* Any major surgery, chemotherapy or immunotherapy within the last 21 days
* Evidence of hepatitis B virus, hepatitis C virus or known HIV infection
* Autologous hematologic stem cell transplant within 3 months of study entry. Prior Allogeneic hematologic stem cell transplant is excluded
* Transformation of CLL to aggressive Non-Hodgkin's Lymphoma (NHL) (Richter's transformation)
* Prior therapy with obinutuzumab and/or chlorambucil or a PI3K delta inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (147):
- United States (103):
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Mobile, Alabama
  - TG Therapeutics Investigational Trial Site, Chandler, Arizona
  - TG Therapeutics Investigational Trial Site, Phoenix, Arizona
  - TG Therapeutics Investigational Trial Site, Tucson, Arizona
  - TG Therapeutics Investigational Trial Site, Fayetteville, Arkansas
  - TG Therapeutics Investigational Trial Site, Concord, California
  - TG Therapeutics Investigational Trial Site, Duarte, California
  - TG Therapeutics Investigational Trial Site, Greenbrae, California
  - TG Therapeutics Investigational Trial Site, Pismo Beach, California
  - TG Therapeutics Investigational Trial Site, Pleasanton, California
  - TG Therapeutics Investigational Trial Site, San Diego, California
  - TG Therapeutics Investigational Trial Site, Santa Barbara, California
  - TG Therapeutics Investigational Trial Site, Whittier, California
  - TG Therapeutics Investigational Trial Site, Aurora, Colorado
  - TG Therapeutics Investigational Trial Site, Denver, Colorado
  - TG Therapeutics Investigational Trial Site, Bridgeport, Connecticut
  - TG Therapeutics Investigational Trial Site, New Haven, Connecticut
  - TG Therapeutics Investigational Trial Site, Stamford, Connecticut
  - TG Therapeutics Investigational Trial Site, Newark, Delaware
  - TG Therapeutics Investigational Trial Site, Boca Raton, Florida
  - TG Therapeutics Investigational Trial Site, Fort Myers, Florida
  - TG Therapeutics Investigational Trial Site, Jacksonville, Florida
  - TG Therapeutics Investigational Trial Site, Ocala, Florida
  - TG Therapeutics Investigational Trial Site, Pensacola, Florida
  - TG Therapeutics Investigational Trial Site, St. Petersburg, Florida
  - TG Therapeutics Investigational Trial Site, Tallahassee, Florida
  - TG Therapeutics Investigational Trial Site, Tampa, Florida
  - TG Therapeutics Investigational Trial Site, West Palm Beach, Florida
  - TG Therapeutics Investigational Trial Site, Albany, Georgia
  - TG Therapeutics Investigational Trial Site, Macon, Georgia
  - TG Therapeutics Investigational Trial Site, Chicago, Illinois
  - TG Therapeutics Investigational Trial Site, Decatur, Illinois
  - TG Therapeutics Investigational Trial Site, Maywood, Illinois
  - TG Therapeutics Investigational Trial Site, Niles, Illinois
  - TG Therapeutics Investigational Trial Site, Peoria, Illinois
  - TG Therapeutics Investigational Trial Site, Swansea, Illinois
  - TG Therapeutics Investigational Trial Site, Urbana, Illinois
  - TG Therapeutics Investigational Trial Site, Fort Wayne, Indiana
  - TG Therapeutics Investigational Trial Site, Indianapolis, Indiana
  - TG Therapeutics Investigational Trial Site, Ames, Iowa
  - TG Therapeutics Investigational Trial Site, Cedar Rapids, Iowa
  - TG Therapeutics Investigational Trial Site, Kansas City, Kansas
  - TG Therapeutics Investigational Trial Site, Westwood, Kansas
  - TG Therapeutics Investigational Trial Site, Louisville, Kentucky
  - TG Therapeutics Investigational Trial Site, Baltimore, Maryland
  - TG Therapeutics Investigational Trial Site, Bethesda, Maryland
  - TG Therapeutics Investigational Trial Site, Columbia, Maryland
  - TG Therapeutics Investigational Trial Site, Boston, Massachusetts
  - TG Therapeutics Investigational Trial Site, Worcester, Massachusetts
  - TG Therapeutics Investigational Trial Site, Ann Arbor, Michigan
  - TG Therapeutics Investigational Trial Site, Detroit, Michigan
  - TG Therapeutics Investigational Trial Site, Jackson, Michigan
  - TG Therapeutics Investigational Trial Site, Saint Louis Park, Minnesota
  - TG Therapeutics Investigational Trial Site, Columbia, Missouri
  - TG Therapeutics Investigational Trial Site, Kansas City, Missouri
  - TG Therapeutics Investigational Trial Site, Lincoln, Nebraska
  - TG Therapeutics Investigational Trial Site, Las Vegas, Nevada
  - TG Therapeutics Investigational Trial Site, Lebanon, New Hampshire
  - TG Therapeutics Investigational Trial Site, Morristown, New Jersey
  - TG Therapeutics Investigational Trial Site, Somerville, New Jersey
  - TG Therapeutics Investigational Trial Site, East Setauket, New York
  - TG Therapeutics Investigational Trial Site, Glens Falls, New York
  - TG Therapeutics Investigational Trial Site, Syracuse, New York
  - TG Therapeutics Investigational Trial Site, Charlotte, North Carolina
  - TG Therapeutics Investigational Trial Site, Durham, North Carolina
  - TG Therapeutics Investigational Trial Site, Hickory, North Carolina
  - TG Therapeutics Investigational Trial Site, Kinston, North Carolina
  - TG Therapeutics Investigational Trial Site, Raleigh, North Carolina
  - TG Therapeutics Investigational Trial Site, Washington, North Carolina
  - TG Therapeutics Investigational Trial Site, Canton, Ohio
  - TG Therapeutics Investigational Trial Site, Cincinnati, Ohio
  - TG Therapeutics Investigational Trial Site, Toledo, Ohio
  - TG Therapeutics Investigational Trial Site, Portland, Oregon
  - TG Therapeutics Investigational Trial Site, Springfield, Oregon
  - TG Therapeutics Investigational Trial Site, Camp Hill, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Danville, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Hershey, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Philadelphia, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Pittsburgh, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Pawtucket, Rhode Island
  - TG Therapeutics Investigational Trial Site, Greenville, South Carolina
  - TG Therapeutics Investigational Trial Site, Sioux Falls, South Dakota
  - TG Therapeutics Investigational Trial Site, Watertown, South Dakota
  - TG Therapeutics Investigational Trial Site, Chattanooga, Tennessee
  - TG Therapeutics Investigational Trial Site, Nashville, Tennessee
  - TG Therapeutics Investigational Trial Site, Austin, Texas
  - TG Therapeutics Investigational Trial Site, Bedford, Texas
  - TG Therapeutics Investigational Trial Site, Fort Worth, Texas
  - TG Therapeutics Investigational Trial Site, Houston, Texas
  - TG Therapeutics Investigational Trial Site, San Antonio, Texas
  - TG Therapeutics Investigational Trial Site, Tyler, Texas
  - TG Therapeutics Investigational Trial Site, Ogden, Utah
  - TG Therapeutics Investigational Trial Site, Blacksburg, Virginia
  - TG Therapeutics Investigational Trial Site, Charlottesville, Virginia
  - TG Therapeutics Investigational Trial Site, Fort Belvoir, Virginia
  - TG Therapeutics Investigational Trial Site, Olympia, Washington
  - TG Therapeutics Investigational Trial Site, Seattle, Washington
  - TG Therapeutics Investigational Trial Site, Spokane, Washington
  - TG Therapeutics Investigational Trial Site, Vancouver, Washington
  - TG Therapeutics Investigational Trial Site, Yakima, Washington
  - TG Therapeutics Investigational Trial Site, Milwaukee, Wisconsin
  - TG Therapeutics Investigational Trial Site, Wauwatosa, Wisconsin
- Israel (7):
  - TG Therapeutics Investigational Trial Site, Ashkelon
  - TG Therapeutics Investigational Trial Site, Beersheba
  - TG Therapeutics Investigational Trial Site, Haifa
  - TG Therapeutics Investigational Trial Site, Jerusalem
  - TG Therapeutics Investigational Trial Site, Nahariya
  - TG Therapeutics Investigational Trial Site, Petah Tikva
  - TG Therapeutics Investigational Trial Site, Tel Aviv
- Italy (5):
  - TG Therapeutics Investigational Trial Site, Bologna
  - TG Therapeutics Investigational Trial Site, Ferrara
  - TG Therapeutics Investigational Trial Site, Milan
  - TG Therapeutics Investigational Trial Site, Rome
  - TG Therapeutics Investigational Trial Site, Torino
- Poland (8):
  - TG Therapeutics Investigational Trial Site, Chorzów
  - TG Therapeutics Investigational Trial Site, Gdynia
  - TG Therapeutics Investigational Trial Site, Krakow
  - TG Therapeutics Investigational Trial Site, Lodz
  - TG Therapeutics Investigational Trial Site, Lublin
  - TG Therapeutics Investigational Trial Site, Słupsk
  - TG Therapeutics Investigational Trial Site, Warsaw
  - TG Therapeutics Investigational Trial Site, Wroclaw
- Russia (9):
  - TG Therapeutics Investigational Trial Site, Krasnozatonskiy
  - TG Therapeutics Investigational Trial Site, Moscow
  - TG Therapeutics Investigational Trial Site, Perm
  - TG Therapeutics Investigational Trial Site, Petrozavodsk
  - TG Therapeutics Investigational Trial Site, Rodionova
  - TG Therapeutics Investigational Trial Site, Saint Petersburg
  - TG Therapeutics Investigational Trial Site, Smolensk
  - TG Therapeutics Investigational Trial Site, Tula
  - TG Therapeutics Investigational Trial Site, Yaroslavl
- Spain (3):
  - TG Therapeutics Investigational Trial Site, Barcelona
  - TG Therapeutics Investigational Trial Site, Madrid
  - TG Therapeutics Investigational Trial Site, Valencia
- United Kingdom (12):
  - TG Therapeutics Investigational Trial Site, Cambridge
  - TG Therapeutics Investigational Trial Site, Cumbria
  - TG Therapeutics Investigational Trial Site, Dudley West
  - TG Therapeutics Investigational Trial Site, London
  - TG Therapeutics Investigational Trial Site, Northbrook
  - TG Therapeutics Investigational Trial Site, Northumbria
  - TG Therapeutics Investigational Trial Site, Norwich
  - TG Therapeutics Investigational Trial Site, Peterborough
  - TG Therapeutics Investigational Trial Site, Southampton
  - TG Therapeutics Investigational Trial Site, St. James
  - TG Therapeutics Investigational Trial Site, Sunderland
  - TG Therapeutics Investigational Trial Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at multiple investigative sites in the United States, Israel, Italy, Poland, Russian Federation, Spain and the United Kingdom from 19 November 2015 to 22 February 2023.
Groups:
- Experimental: Arm A: Ublituximab + Umbralisib: Participants received ublituximab, 150 milligrams (mg), intravenously (IV), on Day 1, 750 mg on Day 2, followed by 900 mg on Days 8 and 15 of Cycle 1 (cycle length=28 days), Day 1 of Cycles 2-6, and once every 3 cycles thereafter, along with umbralisib, 800 mg, orally, once daily during each cycle until disease progression, lack of tolerability, or until the treatment is commercially available or up to 87 months.
- Active Comparator: Arm B: Obinutuzumab + Chlorambucil: Participants received obinutuzumab 100 mg, IV on Day 1, 900 mg on Day 2, followed by 1000 mg on Days 8 and 5 of cycle 1 (cycle length = 28 days), Day 1 of Cycle 2-6 along with chlorambucil 0.5 milligrams per kilogram (mg/kg) tablet orally on Days 1 and 15 once daily during each cycle until disease progression, lack of tolerability, or until the treatment is commercially available or up to 87 months.
- Experimental: Arm C: Ublituximab: Participants received ublituximab, 150 mg, IV, on Day 1, 750 mg on Day 2, followed by 900 mg on Days 8 and 15 of Cycle 1 (cycle length=28 days), Day 1 of Cycles 2-6, and once every 3 cycles thereafter, until disease progression, lack of tolerability, or until the treatment is commercially available or up to 87 months.
- Experimental: Arm D: Umbralisib: Participants received umbralisib, 800 mg tablets, orally, once daily during each cycle (cycle length= 28 days) until removal from study or up to 87 months.
Period: Overall Study
Arm/Group | Experimental: Arm A: Ublituximab + Umbralisib | Active Comparator: Arm B: Obinutuzumab + Chlorambucil | Experimental: Arm C: Ublituximab | Experimental: Arm D: Umbralisib
Started | 210 | 211 | 91 | 91
Safety Population (The safety population included all randomized participants who had received at least one dose of study treatment (ublituximab, TGR-1202, obinutuzumab + chlorambucil, or ublituximab + TGR-1202).) | 206 | 200 | 91 | 86
Completed | 0 | 0 | 0 | 0
Not Completed | 210 | 211 | 91 | 91
Not completed — Adverse Event | 16 | 12 | 7 | 13
Not completed — Death | 29 | 10 | 11 | 11
Not completed — Initiation of Non-protocol Intervention | 5 | 3 | 0 | 0
Not completed — Investigator's Decision | 11 | 15 | 6 | 6
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 2 | 1 | 2
Not completed — Progressive Disease Confirmed by Central Radiology | 75 | 113 | 38 | 43
Not completed — Site Terminated by Sponsor | 29 | 12 | 13 | 5
Not completed — Withdrawal by Subject of Consent or to Discontinue Treatment | 29 | 24 | 6 | 5
Not completed — Reason Not Specified | 3 | 7 | 4 | 5
Not completed — Unknown/Missing | 10 | 13 | 4 | 0
Not completed — Non-Compliance with Study | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all randomized participants, regardless of administration of study treatment (ublituximab, TGR-1202, obinutuzumab + chlorambucil, or ublituximab + TGR-1202).
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Arm A: Ublituximab + Umbralisib | Active Comparator: Arm B: Obinutuzumab + Chlorambucil | Experimental: Arm C: Ublituximab | Experimental: Arm D: Umbralisib | Total
Number analyzed (Participants) | 210 | 211 | 91 | 91 | 603
Age, Continuous [Mean (Full Range); unit: years] | 66.2 [39 to 88] | 67.1 [36 to 91] | 67.6 [40 to 88] | 66.3 [43 to 86] | 66.8 [36 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 67 | 23 | 30 | 195
  Male | 135 | 144 | 68 | 61 | 408
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 2 | 3 | 13
  Not Hispanic or Latino | 193 | 194 | 86 | 83 | 556
  Unknown or Not Reported | 14 | 12 | 3 | 5 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 9 | 6 | 5 | 5 | 25
  White | 189 | 195 | 83 | 82 | 549
  Multiple | 2 | 0 | 0 | 0 | 2
  Other | 1 | 1 | 0 | 2 | 4
  Not Reported | 8 | 7 | 2 | 1 | 18

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Criteria
Description: PFS was defined as the interval from enrollment to the earlier of the first documentation of definitive disease progression (PD) or death from any cause. PD was appearance of new nodes >1.5 centimetres (cm) in the longest diameter (LD) and >1.0 in longest perpendicular diameter (LPD), new or recurrent hepatomegaly or splenomegaly, new or reappearance of an unequivocal extra-nodal lesion, ≥50% increase from the nadir in the sum of products of diameters (SPD) of target lesions, ≥50% increase in the LD of an individual node or extra-nodal mass, splenic/hepatic enlargement of ≥50% from nadir, unequivocal increase in the size of non-target disease, transformation to a more aggressive histology, decrease in platelet count or Hgb, >50% decrease from the highest on-study platelet count, >20 grams per Liter (g/L) decrease from the highest on-study hemoglobin (Hgb).
Time Frame: From enrolment to the earlier of the first documentation of definitive disease progression (PD) or death (Up to 87 months)
Population: The ITT population included all randomized participants, regardless of administration of study treatment (ublituximab, TGR-1202, obinutuzumab + chlorambucil, or ublituximab + TGR-1202).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental: Arm A: Ublituximab + Umbralisib | Active Comparator: Arm B: Obinutuzumab + Chlorambucil | Experimental: Arm C: Ublituximab | Experimental: Arm D: Umbralisib
Number analyzed (Participants) | 210 | 211 | 91 | 91
Months | 33.2 [27.7 to 39.6] | 17.5 [16.6 to 22.6] | 32.9 [19.1 to 45.0] | 22.4 [17.2 to 34.7]

2. Secondary Outcome: Overall Response Rate (ORR) Per iwCLL Criteria
Description: ORR=percent of participants who achieve complete response (CR), complete response with incomplete marrow recovery (CRi), partial response (PR) or nodular partial response (nPR).CR: No evidence of new disease; Absolute lymphocyte count(ALC)<4x10^9/liter(L);Regression of all target nodal masses to ≤1.5cm in LD;Normal spleen,liver size;Regression to normal of all nodal non-target disease and disappearance of all detectable;Non-nodal,non-target disease;Morphologically negative bone marrow;No lymphoid nodules;ANC >1.5x10^9/L,platelets≥100x10^9/L,Hgb≥110 g/L.PR:No evidence of new disease; Response in 2 of following if abnormal at baseline: ALC<4x10^9/L or ≥50% decrease from baseline in sum of products of target nodal lesions;splenomegaly; hepatomegaly;≥50% decrease from baseline in CLL marrow infiltrate/B-lymphoid nodules;response in any 1: ANC>1.5x10^9/L, platelets>100x10^9/L,Hgb>110g/L or ≥50% increase over baseline in any of these.CRi:for CR except with ANC<1000/µL and/or platelets<100.
Time Frame: Up to 87 months
Population: The ITT population included all randomized participants, regardless of administration of study treatment (ublituximab, TGR-1202, obinutuzumab + chlorambucil, or ublituximab + TGR-1202). Percentages are rounded off to the nearest decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Arm A: Ublituximab + Umbralisib | Active Comparator: Arm B: Obinutuzumab + Chlorambucil | Experimental: Arm C: Ublituximab | Experimental: Arm D: Umbralisib
Number analyzed (Participants) | 210 | 211 | 91 | 91
percentage of participants | 83.3 | 68.7 | 42.9 | 61.5

3. Secondary Outcome: Complete Response (CR) Rate
Description: The CR rate is defined as the percentage of participants with a best overall response of complete response (CR) or complete response with incomplete marrow recovery (CRi). CR: No evidence of new disease; Absolute lymphocyte count(ALC)<4x10^9/L; Regression of all target nodal masses to ≤1.5 cm in LD; Normal spleen,liver size; Regression to normal of all nodal non-target disease and disappearance of all detectable; Non-nodal, non-target disease; Morphologically negative bone marrow; No lymphoid nodules; ANC>1.5x10^9/L,platelets≥100x10^9/L,hemoglobin (Hgb)≥110 g/L. CRi was as for CR except with ANC <1000/µL and/or platelets <100,000/µL.
Time Frame: Up to 87 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Arm A: Ublituximab + Umbralisib | Active Comparator: Arm B: Obinutuzumab + Chlorambucil | Experimental: Arm C: Ublituximab | Experimental: Arm D: Umbralisib
Number analyzed (Participants) | 210 | 211 | 91 | 91
percentage of participants | 5.7 | 1.4 | 3.3 | 0

4. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate
Description: MRD negativity rate is defined as the percentage of participants who are MRD negative. If a participant was determined to be MRD negative by peripheral blood, a bone marrow aspirate was obtained to assess MRD in the bone marrow.
Time Frame: From Cycle 6 until Cycle 15 (cycle length=28 days) up to approximately 81.5 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Arm A: Ublituximab + Umbralisib | Active Comparator: Arm B: Obinutuzumab + Chlorambucil | Experimental: Arm C: Ublituximab | Experimental: Arm D: Umbralisib
Number analyzed (Participants) | 210 | 211 | 91 | 91
percentage of participants | 29.0 | 34.6 | 36.3 | 5.5

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the interval from the first documentation of CR, CRi, PR, or nPR to the earlier of the first documentation of definitive disease progression or death from any cause.
Time Frame: From first documentation of response to study treatment till disease progression/death (up to approximately 87 months)
Population: The ITT population included all randomized participants, regardless of administration of study treatment (ublituximab, TGR-1202, obinutuzumab + chlorambucil, or ublituximab + TGR-1202). Overall Number of Participants Analyzed is the number of participants with data available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Arm A: Ublituximab + Umbralisib | Active Comparator: Arm B: Obinutuzumab + Chlorambucil | Experimental: Arm C: Ublituximab | Experimental: Arm D: Umbralisib
Number analyzed (Participants) | 175 | 145 | 39 | 56
months | 32.9 [27.8 to 39.4] | 21.9 [14.6 to 26.6] | 47.5 [40.3 to 57.8] | 29.3 [17.1 to 36.5]

6. Secondary Outcome: Number of Participants Experiencing at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product. An AE does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE is any AE that occur after first dosing of study medication and through the end of the study or through 30 days after the last dose of study treatment, or is considered treatment-related regardless of the start date of the event, or is present before first dosing of study medication but worsens in intensity or the investigator subsequently considers treatment-related.
Time Frame: From first dose of study treatment up to end of study (up to approximately 87 months)
Population: The safety population included all randomized participants who had received at least one dose of study treatment (ublituximab, TGR-1202, obinutuzumab + chlorambucil, or ublituximab + TGR-1202
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Arm A: Ublituximab + Umbralisib | Active Comparator: Arm B: Obinutuzumab + Chlorambucil | Experimental: Arm C: Ublituximab | Experimental: Arm D: Umbralisib
Number analyzed (Participants) | 206 | 200 | 91 | 86
Participants | 205 | 195 | 88 | 86

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to end of study (up to approximately 87 months)
Description: The safety population included all randomized participants who had received at least one dose of study treatment (ublituximab, TGR-1202, obinutuzumab + chlorambucil, or ublituximab + TGR-1202.
Groups:
- Active Comparator: Arm B: Obinutuzumab + Chlorambucil: Participants received Obinutuzumab 100 mg, IV on Day 1, 900 mg on Day 2, followed by 1000 mg on Days 8 and 15 of cycle 1 (cycle length = 28 days), Day 1 of Cycle 2-6 along with Chlorambucil 0.5 milligram per kilogram (mg/kg) tablet orally on Days 1 and 15 once daily during each cycle until disease progression, lack of tolerability, or until the treatment is commercially available or up to 87 months.
Arm/Group | Experimental: Arm A: Ublituximab + Umbralisib | Active Comparator: Arm B: Obinutuzumab + Chlorambucil | Experimental: Arm C: Ublituximab | Experimental: Arm D: Umbralisib
All-Cause Mortality (participants affected / at risk) | 82/206 | 40/200 | 25/91 | 29/86
Serious Adverse Events (participants affected / at risk) | 118/206 | 47/200 | 33/91 | 34/86
Other Adverse Events (participants affected / at risk) | 205/206 | 189/200 | 84/91 | 84/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Arm A: Ublituximab + Umbralisib (N=206) | Active Comparator: Arm B: Obinutuzumab + Chlorambucil (N=200) | Experimental: Arm C: Ublituximab (N=91) | Experimental: Arm D: Umbralisib (N=86)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1 | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 2 | 1
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Adrenal mass (Endocrine disorders) | 0 | 0 | 1 | 0
Exfoliation glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Death (General disorders) | 3 | 1 | 2 | 1
Pyrexia (General disorders) | 2 | 3 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 1 | 0 | 0
Chronic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 21 | 4 | 4 | 0
COVID-19 (Infections and infestations) | 13 | 0 | 4 | 1
COVID-19 pneumonia (Infections and infestations) | 10 | 0 | 8 | 0
Sepsis (Infections and infestations) | 7 | 1 | 4 | 2
Urinary tract infection (Infections and infestations) | 5 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 4 | 3 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 2 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 2 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0
Bordetella infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 0 | 0 | 0
Dientamoeba infection (Infections and infestations) | 1 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Medical device site joint infection (Infections and infestations) | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 1 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0 | 0 | 0
Scrotal infection (Infections and infestations) | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Genitourinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0
Clostridium test positive (Investigations) | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 3 | 3 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 2
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1 | 0 | 0
Intracranial mass (Nervous system disorders) | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Transient aphasia (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 1 | 0 | 0 | 0
Binge drinking (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Vascular compression (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Arm A: Ublituximab + Umbralisib (N=206) | Active Comparator: Arm B: Obinutuzumab + Chlorambucil (N=200) | Experimental: Arm C: Ublituximab (N=91) | Experimental: Arm D: Umbralisib (N=86)
Neutropenia (Blood and lymphatic system disorders) | 70 | 79 | 25 | 15
Anaemia (Blood and lymphatic system disorders) | 29 | 25 | 15 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 21 | 44 | 13 | 7
Vision blurred (Eye disorders) | 14 | 6 | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 118 | 45 | 24 | 54
Nausea (Gastrointestinal disorders) | 105 | 75 | 27 | 34
Constipation (Gastrointestinal disorders) | 38 | 23 | 14 | 12
Vomiting (Gastrointestinal disorders) | 38 | 29 | 9 | 14
Abdominal pain (Gastrointestinal disorders) | 27 | 19 | 9 | 6
Dyspepsia (Gastrointestinal disorders) | 24 | 9 | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 15 | 5 | 1 | 5
Abdominal distension (Gastrointestinal disorders) | 13 | 2 | 5 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 | 5 | 6 | 1
Stomatitis (Gastrointestinal disorders) | 12 | 2 | 0 | 4
Fatigue (General disorders) | 76 | 60 | 28 | 22
Pyrexia (General disorders) | 53 | 38 | 22 | 11
Chills (General disorders) | 52 | 33 | 25 | 12
Oedema peripheral (General disorders) | 39 | 12 | 10 | 9
Asthenia (General disorders) | 25 | 13 | 4 | 4
Pain (General disorders) | 13 | 4 | 3 | 1
Chest discomfort (General disorders) | 12 | 7 | 3 | 0
Influenza like illness (General disorders) | 12 | 9 | 2 | 2
Hypogammaglobulinaemia (Immune system disorders) | 19 | 5 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 48 | 26 | 16 | 18
Pneumonia (Infections and infestations) | 27 | 11 | 10 | 6
Urinary tract infection (Infections and infestations) | 26 | 4 | 10 | 2
Sinusitis (Infections and infestations) | 25 | 7 | 6 | 2
Bronchitis (Infections and infestations) | 20 | 5 | 5 | 4
COVID-19 (Infections and infestations) | 17 | 0 | 6 | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 92 | 49 | 36 | 0
Contusion (Injury, poisoning and procedural complications) | 18 | 9 | 7 | 8
Fall (Injury, poisoning and procedural complications) | 13 | 4 | 6 | 4
Alanine aminotransferase increased (Investigations) | 34 | 9 | 6 | 13
Aspartate aminotransferase increased (Investigations) | 29 | 9 | 6 | 11
Neutrophil count decreased (Investigations) | 28 | 21 | 6 | 6
Platelet count decreased (Investigations) | 21 | 19 | 10 | 4
Weight decreased (Investigations) | 16 | 4 | 4 | 10
Blood creatinine increased (Investigations) | 14 | 10 | 6 | 7
Decreased appetite (Metabolism and nutrition disorders) | 42 | 18 | 6 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 29 | 4 | 2 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 15 | 6 | 3 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 13 | 5 | 5 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 13 | 1 | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 12 | 7 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 | 16 | 16 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 15 | 12 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 11 | 4 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 15 | 10 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 7 | 8 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11 | 3 | 1 | 2
Headache (Nervous system disorders) | 56 | 36 | 18 | 17
Dizziness (Nervous system disorders) | 46 | 19 | 14 | 17
Dysgeusia (Nervous system disorders) | 26 | 3 | 1 | 8
Tremor (Nervous system disorders) | 13 | 3 | 5 | 1
Insomnia (Psychiatric disorders) | 41 | 28 | 12 | 7
Anxiety (Psychiatric disorders) | 24 | 11 | 4 | 5
Depression (Psychiatric disorders) | 11 | 6 | 4 | 4
Pollakiuria (Renal and urinary disorders) | 14 | 5 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 62 | 36 | 18 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 | 34 | 20 | 14
Productive cough (Respiratory, thoracic and mediastinal disorders) | 14 | 3 | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 17 | 3 | 8 | 10
Night sweats (Skin and subcutaneous tissue disorders) | 12 | 6 | 9 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 6 | 3 | 8
Hypertension (Vascular disorders) | 27 | 8 | 9 | 16
Flushing (Vascular disorders) | 16 | 18 | 9 | 2
Hypotension (Vascular disorders) | 13 | 17 | 12 | 3
Atrial fibrillation (Cardiac disorders) | 6 | 3 | 5 | 1
Flatulence (Gastrointestinal disorders) | 9 | 3 | 0 | 8
Colitis (Gastrointestinal disorders) | 7 | 0 | 1 | 6
Gastritis (Gastrointestinal disorders) | 7 | 0 | 0 | 5
Non-cardiac chest pain (General disorders) | 4 | 6 | 6 | 2
Seasonal allergy (Immune system disorders) | 3 | 2 | 6 | 2
Clostridium difficile infection (Infections and infestations) | 2 | 1 | 0 | 5
Herpes zoster (Infections and infestations) | 1 | 1 | 7 | 2
White blood cell count decreased (Investigations) | 10 | 17 | 8 | 0
Blood lactate dehydrogenase increased (Investigations) | 5 | 0 | 5 | 5
Lymphocyte count increased (Investigations) | 3 | 2 | 0 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 10 | 5 | 5 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 6 | 5 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 5 | 2
Paraesthesia (Nervous system disorders) | 9 | 5 | 1 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 7 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 6 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 2 | 1 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 5 | 1 | 5
Hot flush (Vascular disorders) | 9 | 10 | 4 | 4

LIMITATIONS AND CAVEATS:
Due to sponsor's business decision, the clinical trial was terminated by the sponsor prematurely. As such, the study results are reflective of the data captured to the time of study termination and with limited data verification.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT02612311/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT02612311/SAP_001.pdf